CLINICAL TRIAL: NCT05532345
Title: Development and Validation of a Machine Learning Model to Differentiate Drug-induced Liver Injury and Autoimmune Hepatitis
Brief Title: Discrimination of DILI and AIH by Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-P2-263-01
Record Dates: First submitted 2022-08-29; First posted 2022-09-08 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Drug-induced Liver Injury; Autoimmune Hepatitis
Keywords: Artificial intelligence; Differential diagnose
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Development group, retrospectively collecting: The training set includes 80% of the development dataset from Beijing Friendship Hospital (Retrospectively collecting DILI 649 cases and AIH 180 cases in total)
- Validation group, retrospectively collecting: The internal validation group includes 20% of the development dataset from Beijing Friendship Hospital (Retrospectively collecting DILI 649 cases and AIH 180 cases in total).
  External validation groups include Fifth Medical Center of Chinese PLA Medical Center(Retrospectively collecting DILI 585 cases and AIH 400 cases in total), Beijing You'an Hospital (Retrospectively collecting DILI 266 cases and AIH 100 cases in total) and additional seven tertiary hospitals throughout China (Retrospectively collecting DILI 182 cases and AIH 92 cases in total, including Tianjin Second People's Hospital, Heilongjiang Provincial Hospital, Affiliated Hospital of Qingdao University, the First Affiliated Hospital of Xiamen University, Traditional Chinese Medical Hospital of Xinjiang Uygur Autonomous Region, Lanzhou University Second Hospital, Qinghai Provincial People's Hospital).
- Real-World validation group, prospectively and retrospectively collecting: Real-World validation data will be prospectively and retrospectively collected from Beijing Friendship Hospital (78 cases for DILI and 51 cases for AIH)

SUMMARY:
A retrospective, multi-center, non-interventional cohort study has been going to explore whether artificial intelligence can discriminate Drug-induced liver injury and Autoimmune hepatitis.

A machine learning-based tool will be developed and validated to help clinicians to differentiate between Drug-induced liver injury and Autoimmune hepatitis

DETAILED DESCRIPTION:
Research Objectives:

1. To develop a machine learning-based model from retrospective data.
2. To validate the machine learning-based model from internal dataset and external datasets nationwide.
3. To setup a website or application based on the above model to discriminate Drug-induced liver injury and Autoimmune hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Drug-induced liver injury

  1. RUCAM ≥6 and met one of the following biochemical conditions: a.) ALT≥5 ULN, b.) or ALP ≥2 ULN, iii) or ALT≥3 ULN and TBil≥2 ULN.
  2. RUCAM was between 3-5, the medical records were further reviewed by the three authors to determine the eligibility.
* Autoimmune hepatitis

  1. The revised International Autoimmune Hepatitis Group (IAIHG) diagnostic score≥6 points.
  2. Liver biopsy available, which is compatible with typical features of AIH.
  3. If liver biopsy was unavailable, patients who achieved biochemical resolution after sustained immunosuppressive therapy.

Exclusion Criteria:

* Drug-induced liver injury

  1. Hepatotropic viral infection: hepatitis A, B, C, D and E.
  2. Non-hepatotropic viral infection: cytomegalovirus (CMV) and Epstein-Barr virus (EBV), etc.
  3. Hypoxic ischemic hepatitis and congestive liver disease.
  4. Alcohol consumption: male >40g/d, female >20g/d, and ≥5 years.
  5. Biliary obstruction, primary biliary cholangitis; primary sclerosing cholangitis.
  6. Autoimmune hepatitis.
  7. Parasitic infection.
  8. Sepsis.
  9. Previous liver transplantation or bone marrow transplantation.
  10. Pregnancy or lactation.
  11. Genetic and metabolic liver diseases.
* Autoimmune hepatitis

  1. Hepatotropic viral infection: hepatitis A, B, C, D and E.
  2. Non-hepatotropic viral infection: cytomegalovirus (CMV) and Epstein-Barr virus (EBV), etc.
  3. Hypoxic ischemic hepatitis and congestive liver disease.
  4. Alcohol consumption: male >40g/d, female >20g/d, and ≥5 years.
  5. Biliary obstruction, primary biliary cholangitis; primary sclerosing cholangitis.
  6. Drug-induced liver injury.
  7. Parasitic infection.
  8. Sepsis.
  9. Previous liver transplantation or bone marrow transplantation.
  10. Pregnancy or lactation.
  11. Genetic and metabolic liver diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with a definite diagnosis of DILI and AIH were recruited from all hospitals between January 2009 to October 2022. This study was approved by the Institutional Ethical Review Board (2022-P2-263-01).
Sampling Method: Non-Probability Sample
Enrollment: 2583 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of the model in the differential diagnosis of DILI and AIH | May 31, 2023
  The ratio of the correct number of forecasts to the total number of forecasts
The confidence of the model in the differential diagnosis of DILI and AIH | May 31, 2023
  The confidence and 95% confidence internal of the model in determining whether each case is DILI or AIH

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan Zhao, Dr., Study Chair — Beijing Friendship Hospital; Ying Sun, Dr., Principal Investigator — The Fifth Medical Department of the PLA; Jing Zhang, Dr., Principal Investigator — Capital Medical University Affiliated Beijing You'an Hospital; Jia Li, Dr., Principal Investigator — Tianjin Second People's Hospital; Liang Wang, Dr., Principal Investigator — Lanzhou University Affiliated Second Hospital; Xiaoli Hu, Dr., Principal Investigator — Heilongjiang provincial hospital; Jingshou Chen, Dr., Principal Investigator — The First Affiliated Hospital of Xiamen University; Feng Guo, Dr., Principal Investigator — Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine; Pingying Li, Dr., Principal Investigator — Qinghai People's Hospital; Qiuju Tian, Dr., Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Wang Y, Lin X, Sun Y, Liu J, Li J, Tian Q, Guo F, Hu X, Wang L, Li P, Chen J, Wang Y, Ma Z, Jia J, Zhang J, Zou Z, Zhao X. Development and Validation of a Novel Model to Discriminate Idiosyncratic Drug-Induced Liver Injury and Autoimmune Hepatitis. Liver Int. 2025 Feb;45(2):e16239. doi: 10.1111/liv.16239. PMID 39817622